CLINICAL TRIAL: NCT04867902
Title: Gaining Optimism After Weight Loss Surgery (GOALS) I: Proof-of-Concept Trial of a Positive Psychology-based Intervention to Increase Physical Activity After Bariatric Surgery
Brief Title: Gaining Optimism After Weight Loss Surgery (GOALS) I
Acronym: GOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emily Feig, Ph.D., Instructor in Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P001006a; 5K23HL148017 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery
Keywords: Positive Psychology; Motivational Interviewing; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Psychology-Motivational Interviewing Intervention (Experimental): Participants will receive a written treatment manual with detailed information about each topic. The intervention consists of 10 weekly phone sessions (30 minutes each). Each session includes a new psychological skill designed to increase positive emotions experienced during physical activity, a motivational skill designed to boost physical activity, and setting a physical activity goal for the next week using information from the Fitbit. A motivational interviewing approach will be used for all topics.
  Interventions: Behavioral: Positive Psychology-Motivational Interviewing Intervention

INTERVENTIONS:
Behavioral: Positive Psychology-Motivational Interviewing Intervention — Participants will receive a written treatment manual with detailed information about each topic. The intervention consists of 10 weekly phone sessions (30 minutes each). Each session includes a new psychological skill designed to increase positive emotions experienced during physical activity, a motivational skill designed to boost physical activity, and setting a physical activity goal for the next week using information from the Fitbit. A motivational interviewing approach will be used for all topics.

SUMMARY:
This study examines the feasibility, acceptability, and preliminary impact of an adapted positive psychology-motivational interviewing (PP-MI) intervention for physical activity among patients who have recently undergone bariatric surgery.

DETAILED DESCRIPTION:
This study will test a positive psychology-motivational interviewing (PP-MI) intervention for physical activity promotion in patients who have had bariatric surgery within the past 6-12 months. The investigators will enroll 12 participants. Study participation includes attending three study visits (two at baseline, one after the intervention) and receiving a 10-week physical activity intervention that includes once-weekly phone calls, a written manual, and a Fitbit activity tracker. Primary outcomes are feasibility and acceptability of the intervention and study procedures. Secondary outcomes include pre-post changes in physical activity and other psychological, behavioral, and physiological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+)
* History of bariatric surgery (gastric bypass or sleeve gastrectomy) at one of two academic medical centers within the past 6-12 months
* Interest in increasing physical activity
* Low physical activity, defined as <200 minutes/week self-reported moderate- to-vigorous physical activity
* Access to telephone for study sessions
* Able to read and speak English

Exclusion Criteria:

* Cognitive deficits precluding participation or informed consent
* Illness likely to lead to death in the next 6 months
* Inability to be physically active (e.g., severe arthritis)
* Participation in another program targeting physical activity besides their standard offerings at the surgery center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily H Feig, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Started | 12
Completed | 8
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Intervention Sessions Completed
Description: Feasibility will be measured by examining the number of completed intervention sessions. The intervention will be considered feasible if at least 7/10 sessions are completed, on average.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
sessions | 8.5 (10)

2. Primary Outcome: Ease and Utility of Intervention Sessions
Description: Acceptability will be measured with ratings of ease and utility after each exercise, measured on a 10-point Likert scale (1=very difficult/not at all helpful, 10=very easy/very helpful). The intervention will be considered acceptable if average ease and utility ratings are at least 7/10.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 range)
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
units on a scale (0-10 range)
  Positive psychology ease | 8.3 (1.6)
  Positive psychology utility | 8.7 (1.4)
  Motivational interviewing ease | 8.8 (1.6)
  Motivational interviewing utility | 8.7 (1.4)

3. Secondary Outcome: Change in Moderate to Vigorous Physical Activity (MVPA)
Description: We will use ActiGraph GT3X-BT accelerometers to objectively measure physical activity for 1 week at each assessment. MVPA will be measured in minutes/week.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 8 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
minutes/week
  Baseline | 105.0 (138.5)
  Follow-up: number analyzed (Participants) | 8
  Follow-up | 223.4 (352.2)

4. Secondary Outcome: Change in Steps
Description: Measured by Actigraph accelerometer, in number of steps per day.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 8 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
steps/day
  Baseline | 5008.8 (6544.9)
  Follow-up: number analyzed (Participants) | 8
  Follow-up | 6544.9 (6303.0)

5. Secondary Outcome: Change in Light Physical Activity
Description: Measured by Actigraph accelerometer, in minutes per week.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 8 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
minutes/week
  Baseline | 1767.6 (339.0)
  Follow-up: number analyzed (Participants) | 8
  Follow-up | 1786.5 (623.5)

6. Secondary Outcome: Change in Sedentary Time
Description: Measured by Actigraph accelerometer, in minutes per day.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 8 participants provided follow-up data
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 11
minutes/day
  Baseline | 691.63 (190.11)
  Follow-up: number analyzed (Participants) | 8
  Follow-up | 743.71 (185.94)

7. Secondary Outcome: Change in Optimism
Description: The Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 11.3 (1.5)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 11.4 (1.8)

8. Secondary Outcome: Change in Depressive Symptoms
Description: The Hospital Anxiety and Depression Scale (HADS)-depression subscale will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 5.0 (4.7)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 3.0 (4.1)

9. Secondary Outcome: Change in Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 7.5 (4.2)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 4.7 (4.6)

10. Secondary Outcome: Change in Motivation to Change
Description: The University of Rhode Island Change Assessment (URICA) is a well-validated, 32-item measure that will be used to assess motivation to change. Higher scores indicate higher motivation to change. Scores range from -2 to 14.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 10.39 (1.12)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 10.36 (1.45)

11. Secondary Outcome: Change in Exercise Identity
Description: The Exercise Identity Scale (EIS) is a well-validated, 9-item measure that will be used to assess the extent to which exercise contributes to one's role-identity (Range: 9-63). Higher scores indicate stronger exercise identity.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 26.6 (8.3)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 39.9 (11.4)

12. Secondary Outcome: Change in General Self-Efficacy
Description: Self-efficacy will be measured using the General Self Efficacy scale (GSE), a validated measure of self-efficacy, given its links to improved adherence. Higher scores indicate greater self-efficacy. Possible scores range from 10-40.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 32.5 (3.6)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 34.6 (1.8)

13. Secondary Outcome: Change in Exercise-specific Self-efficacy
Description: Exercise-specific self-efficacy will be measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assesses self-efficacy for exercise (Range: 0-90). Higher scores indicate higher self-efficacy.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 44.6 (19.1)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 55.3 (15.6)

14. Secondary Outcome: Change in Internalized Weight Bias
Description: The Weight Bias Internalization Scale - Modified (WBIS-M) is a well-validated, 11-item measure that will be used to measure internalized weight bias (Range: 11-77). Higher scores indicate greater internalized weight bias.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 4.0 (1.6)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 3.2 (1.9)

15. Secondary Outcome: Change in Body Image
Description: Body image will be assessed using the Multidimensional Body-Self Relations Questionnaire (MBSRQ) Appearance Evaluation subscale. Higher scores indicate better body image and possible scores range from 1-5.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 2.42 (1.06)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 3.26 (1.10)

16. Secondary Outcome: Change in Bariatric Surgery-specific Diet and Vitamin Adherence
Description: The Bariatric Surgery Self-Management Questionnaire (BSSQ) is a validated measure that will be used to assess adherence to diet and vitamin recommendations after bariatric surgery. Higher scores indicate better adherence to diet and vitamin recommendations. Possible scores range from 0-66.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 7 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 41.7 (8.0)
  Follow-up: number analyzed (Participants) | 7
  Follow-up | 46.0 (5.0)

17. Secondary Outcome: Change in Self-Reported Physical Activity
Description: The International Physical Activity Questionnaire (IPAQ) - Short Form is a well-validated 7-day physical activity recall assessment for physical activity. Activity will be measured by the number of minutes per day of moderate or greater activity per week.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 8 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
minutes/day
  Baseline | 11.25 (13.41)
  Follow-up | 44.02 (56.01)

18. Secondary Outcome: Change in Body Weight
Description: Body weight (in pounds) will be measured on a calibrated scale.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
pounds
  Baseline | 257.95 (146.65)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 199.83 (36.04)

19. Secondary Outcome: Change in Waist Circumference (in Centimeters)
Description: Waist circumference will be measured by a nurse.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
cm
  Baseline | 114.4 (27.5)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 102.2 (14.1)

20. Secondary Outcome: Change in Systolic Blood Pressure
Description: Blood pressure will be measured by a nurse in mmHG.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
mmHG
  Baseline | 116.83 (16.03)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 117.83 (10.01)

21. Secondary Outcome: Change in Aerobic Capacity and Endurance
Description: The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
meters
  Baseline | 494.7 (81.1)
  Follow-up | 583.2 (62.3)

22. Secondary Outcome: Change in Social Support for Exercise
Description: The Social Support and Exercise Survey is a 13-item validated measure that assesses social support for exercising from family and friends over the past 3 months. Scores range from 20 to 200, with higher scores indicating more social support.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 42.92 (14.18)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 54.33 (12.61)

23. Secondary Outcome: Change in Social Support for Eating Habits - Encouragement Subscale
Description: The Social Support and Eating Habits Survey encouragement subscale is a 5-item validated measure that assesses social support for healthy eating from family and friends over the past 3 months. Scores range from 10 to 80, with higher scores indicating more social support.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
score on a scale
  Baseline | 24.92 (10.52)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 26.17 (6.18)

24. Secondary Outcome: Change in Body Composition
Description: The measurement of body fat in relation to lean body mass will be measured using bio-electrical impedance.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
percentage of body fat
  Baseline | 40.1 (13.3)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 39.1 (13.5)

25. Secondary Outcome: Change in A1C
Description: Hemoglobin A1C will be measured via blood draw. A higher percentage means higher blood glucose values.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
percentage of glycosylated hemoglobin
  Baseline | 5.19 (0.38)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 5.25 (0.35)

26. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: HDL will be measured via blood draw. Higher levels of HDL in the blood means better absorption and clearing of cholesterol.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
mg/dL
  Baseline | 50.58 (9.18)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 56.33 (11.76)

27. Secondary Outcome: Change in Inflammation
Description: C-reactive protein will be measured via blood draw as a measure of inflammation in mg/dL.
Time Frame: Baseline and 10-Week Follow-Up
Population: Only 6 participants provided follow-up data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
Number analyzed (Participants) | 12
mg/dL
  Baseline | 3.47 (3.33)
  Follow-up: number analyzed (Participants) | 6
  Follow-up | 4.17 (3.59)

ADVERSE EVENTS:
Time Frame: During each participant's study participation (approximately 14 weeks).
Arm/Group | Positive Psychology-Motivational Interviewing Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04867902/Prot_SAP_000.pdf